CLINICAL TRIAL: NCT04047043
Title: Evaluation of Serum Taurine as a Prognostic Marker for Graft Function in Adult Egyptian Patients Undergoing Living Donor Liver Transplant : A Prospective Study
Brief Title: Evaluation of Serum Taurine as a Prognostic Marker for Graft Function in Adult Egyptian Patients Undergoing Living Donor Liver Transplant
Acronym: Taurine/LDLT
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Assistant Professor, Ain Shams University
Other Study IDs: IRB 0006379
Record Dates: First submitted 2019-07-31; First posted 2019-08-06 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Taurine
Keywords: Taurine/graft function/LDLT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Taurine > 30 μmol/L: serum taurine level
  Interventions: Diagnostic Test: serum taurine
- Taurine 30-20 μmol/L: serum taurine level
  Interventions: Diagnostic Test: serum taurine
- Taurine < 20 μmol/L: serum taurine level
  Interventions: Diagnostic Test: serum taurine

INTERVENTIONS:
Diagnostic Test: serum taurine — blood sample for serum taurine level

SUMMARY:
Although the hepatoprotective properties of taurine are well established, however the correlation of the perioperative serum level of this amino acid in the recipients of living donor liver transplantation ( LDLT ) and graft function has not been investigated so far. In the present study, we proposed to examine the serum taurine as a prognostic marker for graft function in adult Egyptian patients undergoing LDLT

DETAILED DESCRIPTION:
* All selected adult patients undergoing LDLT will be admitted to the ICU post LDLT
* Preoperative assessment and preparation will be done according to the standard protocol of the hospital. After full clinical examinations using MELD score corrected for serum sodium level ), imaging techniques (Abdominal U.S; abdominal triphasic CAT Scan, liver biopsy, CT volumetry, upper and lower GIT endoscopy, CT chest, bone scan in HCC patients, renal scan in patients with urinary creatinine clearance < 60 ml/min), pulmonary function test, carotid duplex and dobutamine ECHO will be done for all recipients .
* Serum level of AST, ALT, bilirubin, albumin, ALP, GGT, prothrombin, INR, partial thrombin time, factor V, fasting blood glucose, CBC, CRP, Procalcitonin, urea, creatinine, urinary creatinine clearance, serum electrolytes, urine and stool analysis will be done for all patients.
* Analysis of serum levels of specific liver tumor markers including AFP, beside taurine as a possible new marker will be done for all patients .
* HCV and HBV will be detected for all patients by PCR technique.
* CMV IgM , EBV IgM ,HSV IgM will be done for all patients.
* After 12 hours fasting, 10 ml of venous blood will be collected, in plain tube and allowed to clot for 1/2 an hour. Then, it will be centrifuged at 3,000 rpm for 10 min. The serum will be separated and stored at -20 Cº to avoid loss of biological activity until the batch analysis for serum taurine which will be measured four times for the recipient ( preoperative before induction of anesthesia , 7, 14 days and 30 days post transplant ) by high performance liquid chromatography (HPLC) .

Recipient patients will be divided into 3 groups according to preoperative serum taurine .

* Group 1 ( > 30 μmol/L) (20 cases)
* Group 2 (30-20 μmol/L) (20 cases)
* Group 3 (< 20 μmol/L ) (20 cases)

Intraoperatively, both standard anesthetic and piggyback techniques for hepatic transplantation will be performed by the same anesthesia and surgical team who will be blinded to study medication. Intraoperative blood loss, graft weight, graft weight to recipient weight ratio (GWRWR), blood products transfused, and intraoperative adverse events will be recorded. At the end of surgery, patients will be transferred to the ICU and will be monitored and receive the standard protocol for postoperative management after liver transplantation .

All patients will be assessed for primary graft function (PGF) on a daily basis during the first week post-transplant. Primary graft dysfunction includes one or more of the following variables: (1) bilirubin ≥10 mg/dL on postoperative day 7; (2) INR ≥1.6 on postoperative day 7; and (3) ALT or AST >2000 IU/L within 7 postoperative days.

The primary outcome include correlation between serum taurine levels ( μmol/L) of recipients and graft function which will be detected by liver profile. Secondary outcomes include 30 days mortality (days), the duration of ICU and hospital stays (days) and any recorded post operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Recipient age ≥18 years.
* Donor age between 18 and 45 years
* ABO group compatibility with the recipient
* Normal psychological workup.

Exclusion Criteria:

* Recipients patients with pre-existing renal failure requiring hemodialysis or continuous hemofiltration, glomerular filtration rate ≤ 30 ml /min by renal scan, ..
* Re-transplant
* HA1C > 7%
* Pregnancy.
* Donors with fatty liver.
* Estimated remnant liver volume for donor is < 30% of total liver volume.
* Donor body mass index > 28 kg/m².
* Donor with abnormal biliary anatomy.
* Donor with steatosis > 10%.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After reviewing of literature, no previous similar research was done before to study the effect of recipient serum taurine on graft survival after living donor liver transplant). So considering an exploratory study, the study will include 20 cases with taurine >30 μmol/L, 20 cases with taurine 20-30 μmol/L and 20 cases with taurine <20 μmol/L (60 total).
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Taurine level in micro mol/L | 7 months
  Taurine level preoperative, 7th,14 th and 30 days post liver transplantation will be assesd and correlated with graft function

SECONDARY OUTCOMES:
Seventh day syndrome, 30 days mortality (days), the duration of ICU and hospital stays (days). | 7 months
  Taurine level will be correlated with these parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa El Gendy, Cairo, Ain Shams University Specialized Hospital, Egypt

IPD SHARING:
Plan to Share IPD: Undecided